CLINICAL TRIAL: NCT00733837
Title: Cervical Multifidus Muscle Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Logan College of Chiropractic (Other)
Responsible Party: Kristan Giggey, DC, Logan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RD0627080141
Record Dates: First submitted 2008-08-11; First posted 2008-08-13 (Estimated); Last update posted 2008-12-18 (Estimated); Status verified 2008-12

CONDITIONS: Proprioception; Muscle Activation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): This is a repeated measures study. All participants experience the same conditions.
  Interventions: Other: Nonspecific, Innocuous, Mechanoreceptor Stimulation

INTERVENTIONS:
Other: Nonspecific, Innocuous, Mechanoreceptor Stimulation — A custom device will be used to provide light manual cervical traction

SUMMARY:
The purpose of this study is to determine the relationship between cervical multifidi thickness, cervical spine proprioception and possible reflex activation of cervical multifidi through stimulation of joint mechanoreceptors. Cervical mechanoreceptors will be activated with an innocuous, nonspecific stimulation. Participants will have cervical spine proprioception assessed through joint position sense testing. The multifidus muscle thickness and activation state is to be assessed by sonography. These measures are done pre & post to the innocuous stimulation. There is no specific hypothesis.

ELIGIBILITY:
Inclusion Criteria:

* Logan student, staff, or faculty, ages 18 - 30 years

Exclusion Criteria:

* Fractures
* Tumors
* Dislocations
* Myopathies
* Signs and/or symptoms of neuromotor disorders
* Consumption of prescription drugs that affect the nervous system
* Recent cervical spine injuries or surgeries
* Pain
* Manipulative therapy within the preceding 7 days
* Neck pain

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-07; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
sonographic measurement of multifitus thickness | pre - post

SECONDARY OUTCOMES:
cervical spine repositioning error | pre - post

CONTACTS AND LOCATIONS:
Locations (1):
- Logan College, Chesterfield, Missouri, United States